CLINICAL TRIAL: NCT06757296
Title: Endoscopic Conversion of Sleeve Gastrectomy to Single Anastomosis Sleeve-ileal Bypass (SASI) for Gastroesophageal Reflux (GERD), Primary and Secondary Non-responder.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore Health Services (Other)
Collaborators: Changi General Hospital (Other); Sengkang General Hospital (Other)
Responsible Party: Principal Investigator, Chin Hong Lim, Doctor, Singapore Health Services
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-3067
Record Dates: First submitted 2024-01-19; First posted 2025-01-03 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2024-12

CONDITIONS: Metabolic Syndrome; Severe Obesity; Reflux, Gastroesophageal; Bariatric Surgery
Keywords: SASI; Severe Obesity; Bariatric Surgery
MeSH Terms: conditions — Metabolic Syndrome; Obesity, Morbid; Gastroesophageal Reflux

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (Experimental): Endoscopic SASI
  Interventions: Procedure: Endoscopic SASI

INTERVENTIONS:
Procedure: Endoscopic SASI — Endoscopic conversion to sleeve gastrectomy to SASI

SUMMARY:
The aim of this study is to determine the feasibility and effectiveness of endoscopic anastomosis of sleeve gastrectomy to ileum with a lumen apposing metal stent (LAMS) after a failed sleeve gastrectomy.

DETAILED DESCRIPTION:
The current standard of care for patients who experience insufficient weight loss, weight re-gain or Type II diabetes relapse after a sleeve gastrectomy is a revisional laparoscopic sleeve gastrectomy.

However, such revisional procedure is commonly associated with high mortality and morbidity due to protein malnutrition. A noval bariatric procedure, single anastomosis sleeve ileal (SASI) bypass has emerged recently.

In this study, we are utilizing an incisionless novel endoscopic technique to efficiently replicate the anatomical features and physiological effects of SASI.

ELIGIBILITY:
Inclusion Criteria:

Subject must meet all the inclusion criteria to participate in this study and list each criterion.

1. Age: 21-65 years
2. Patients going for LSG at participating hospitals.
3. Able to provide informed consent

Individuals below age 21 would not be recruited as this is a study in the adult population. Individuals above age 65 are excluded to minimize the procedure risk.

Exclusion Criteria:

1. Patients who were breast feeding or pregnant
2. Severe psychiatric illness
3. Eating disorder
4. Active neoplastic disease
5. End-stage renal disease
6. Patients with bleeding diathesis
7. Patients with pacemakers or implantable cardiac defibrillators
8. Significant cardiovascular disease (e.g., acute myocardial infarction, congestive cardiac failure, ischemic heart disease, atrial fibrillation, sick sinus syndrome, supraventricular tachycardia)
9. Any factors likely to limit adherence to study protocol (e.g., dementia; alcohol or substance abuse; history of unreliability in medication taking or appointment keeping; significant concerns about participation in the study from spouse, significant other or family members)
10. Treatment with anti-platelet agents that could not be temporarily discontinued

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2025-02-03 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Total amount of weight loss | 6 months
  Amount of weight loss after endoscopic conversion to SASI will be measured in kg and will be reported in percentage (%).

SECONDARY OUTCOMES:
HbA1c | 6 months
  HbA1c levels will be measured and reported in percentage (%)
GERD symptoms | 6 months
  Quality of Life in Reflux And Dyspepsia (QoLRAD) is a questionnaire used to assess how gastroesophageal reflux disease (GERD) and dyspepsia (indigestion) affects a person's quality of life.
  The total score will be calculated from the questionnaire and a reduction in QoLRAD score over time will demonstrate improvement.

OTHER OUTCOMES:
Feasibility & Safety | 30 days
  Technical success rate & procedure related complications.
  Number of adverse events will be recorded at all times to determine the feasibility and safety of the study procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Chin Hong Lim, MD, Principal Investigator — Singapore General Hospital
Locations (3):
- Singapore (3):
  - Changi General Hospital, Singapore
  - Sengkang General Hospital, Singapore
  - Singapore General Hospital, Singapore

IPD SHARING:
Plan to Share IPD: No